CLINICAL TRIAL: NCT00784082
Title: Inflammatory Response to Hydroxyurea Therapy in Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P080102; 2008-005077-35 (EudraCT Number)
Record Dates: First submitted 2008-10-27; First posted 2008-11-03 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Sickle Cell Disease
Keywords: Sickle cell disease, hydroxyurea, inflammation
MeSH Terms: conditions — Anemia, Sickle Cell; Inflammation | interventions — Hydroxyurea; Pharmaceutical Preparations

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — Sample with DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Homozygous SS sickle cell children: Hydroxycarbamide, Hydroxyurea (drug):
  1. Homozygous SS sickle cell children, aged > 3 years, of sub-Saharian Africa extraction, in a steady-state of disease , taken no drug except penicillin-V, folate or iron supplementation, hydroxyurea, divided into three groups :
     * children treated with hydroxyurea 20-25 mg/kg/day since at least 3 months with clinical efficacy on vaso-occlusive events
     * untreated children with major vaso-occlusive events
     * children > 5 year-old without a history of vaso-occlusive events
  2. Controls : heterozygous AS parents or siblings of the patients, and AA siblings or healthy African unrelated subjects, aged > 3 years, taken no drug on the day of blood sampling.
  Interventions: Drug: Hydroxycarbamide, Hydroxyurea (drug)
- Homozygous SS children: Hydroxycarbamide, Hydroxyurea (drug):
  1. Homozygous SS children, aged > 3 years, of sub-Saharian Africa extraction, in a steady-state of disease, taken no drug except penicillin-V, folate or iron supplementation, hydroxyurea, divided into three groups :
     * children treated with hydroxyurea 20-25 mg/kg/day since at least 3 months with clinical efficacy on vaso-occlusive events
     * untreated children with major vaso-occlusive events
     * children > 5 year-old without a history of vaso-occlusive events
  2. Controls : heterozygous AS parents or siblings of the patients, and AA siblings or healthy African unrelated subjects, aged > 3 years, taken no drug on the day of blood sampling.
  Interventions: Drug: Hydroxycarbamide, Hydroxyurea (drug)

INTERVENTIONS:
Drug: Hydroxycarbamide, Hydroxyurea (drug) — hydroxyurea 20-25 mg/kg/day since at least 3 months

SUMMARY:
In sickle cell disease (SCD), polymerisation of haemoglobin S and the resulting shape change of the red blood cells (RBC) lead to vascular occlusion and severe painful crises. Permanent inflammatory state and abnormal RBC adhesion to the endothelium trigger these phenomenon. Hydroxyurea (HU) is the only drug that has been shown to reduce clinical severity of SCD, and this was initially attributed to the stimulation of foetal haemoglobin (HbF). However, the clinical response does not correlate consistently with the degree and time of HbF increment, suggesting that HU clinical benefits may involve other mechanisms such as the induction of natural anti-inflammatory response via the hypothalami-pituitary-adrenal axis.

DETAILED DESCRIPTION:
Plasmatic proinflammatory molecules (C-reactive protein, orosomucoid, RANTES, IL-6, IL-8, MCP-1, IL-1A, IL-1B, ET-1, IL-4, IL-10, TNFalpha, IFNgamma), hormones from the hypothalami-pituitary-adrenal axis (cortisol, ACTH), and hypothalamic peptids (arginine vasopressin, corticotrophin-releasing hormone) will be measured from SCD children treated or not with HU (20 treated children, 20 untreated children with a history of vaso-occlusive events, 20 asymptomatic children, and 20 healthy African controls).

ELIGIBILITY:
INCLUSION CRITERIA:

1. Homozygous SS sickle cell children, aged > 3 years, of sub-Saharian Africa extraction, in a steady-state of disease (free of any infectious or vaso-occlusive events for the 4 weeks prior to and 2 weeks after blood sampling, and transfusion-free for 4 months prior to blood sampling), taken no drug except penicillin-V, folate or iron supplementation, hydroxyurea, divided into three groups :

   * children treated with hydroxyurea 20-25 mg/kg/day since at least 3 months with clinical efficacy on vaso-occlusive events
   * untreated children with major vaso-occlusive events
   * children > 5 year-old without a history of vaso-occlusive events Signed informed consent obtained from the subjects (if possible) and their parents
2. Controls : heterozygous AS parents or siblings of the patients, and AA siblings or healthy African unrelated subjects, aged > 3 years, taken no drug on the day of blood sampling.

Signed informed consent obtained from the subjects (if possible) and their parents

EXCLUSION CRITERIA:

* Children in a acute-phase of the disease
* Parent's or patient's refusal
* Taking any drug except penicillin-V, folate or iron supplementation, hydroxyurea
* Un-healthy control or taking drug

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Homozygous SS sickle cell children, aged > 3 years, of sub-Saharian Africa heterozygous AS parents or siblings of the patients, and AA siblings or healthy African unrelated subjects, aged > 3 years
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2009-05; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Determination of plasma inflammatory markers | Day 1
  Determination of plasma inflammatory markers (RANTES, IL-6, IL-8, MCP-1, IL-1A, IL-1B, ET-1, IL-4, IL-10, TNF a,, IFN g) of hormones of the pituitary-adrenal (cortisol, ACTH) and hypothalamic peptides (AVP, CRH).

SECONDARY OUTCOMES:
Clinical data | Day 1
  Clinical data (age, sex of the patient and his parent or siblings, frequency of painful crises requiring hospitalization, measured / year in the three years prior to the study, frequency and causes acute anemic episodes, whether or not a hepatosplenomegaly)
Hematological at baseline | Day 1
  Hematological at baseline (Hb, reticulocytes, MCV, platelets, leukocytes, PN and monocytes, lymphocytes, erythroblasts, iron status)
Determination of HbF | Day 1
  Determination of HbF
Determination of markers of the "acute phase" | Day 1
  Determination of markers of the "acute phase": CRP and orosomucoid
Plasma concentrations | Day 1
  Plasma concentrations of HU just before taking HU (residual) and H2 after dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Hélène Odièvre, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Louis Mourier, Colombes, France